CLINICAL TRIAL: NCT03074188
Title: Prevalence of Oral Findings in Adult Patients With Chronic Kidney Disease "Cross Sectional
Brief Title: Prevalence of Oral Findings in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alaa Mostafa Hassan Elnaggar (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Alaa Mostafa Hassan Elnaggar, internal resident at oral medicine department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: kidney _oral findings
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Oral Disease; Chronic Kidney Diseases
Keywords: oral findings or oral manifestation; pre-dialysis stage or end stage renal disease
MeSH Terms: conditions — Mouth Diseases; Renal Insufficiency, Chronic; Oral Manifestations; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- pre-dialysis patients
- end stage renal disease

SUMMARY:
There are severe deficiency of database concerning the oral health status in both pre-dialysis and end stage renal disease in Egyptian population. Our aim in the present study is to assess the oral health of the chronic kidney disease patients to increase their awareness and minimize all the possible risk factors, to achieve a proper management for all oral problems.

DETAILED DESCRIPTION:
The study will be held in the Nephrology units at the Kasr Al-Ainy Cairo university hospital. The data collected through the questionnaire will be obtained through an interview between the investigator and the patient. Clinical examination will be performed for both oral (soft tissue) and dental (hard) tissue. For patients undergoing dialysis, examination will be performed before dialysis therapy.

Selection bias: will be minimized by enrolling the participants in the study in a consecutive order of the entering the clinic.

Non-respondent bias: will be minimized by explaining to the participants the aim of the study and their importance and role in the study.

Incomplete records: will be excluded from statistical analysis with reporting the cause of not completing the record.

Sample size estimation:

Using a precision of 5, a design effect set at 1 with 90% CI (confidence interval), a total sample size of 250 pre-dialysis patients and 200 end stage renal disease patients will be sufficient. The sample size was calculated by Epi info software.

The sample will be divided between two researchers; each researcher will have 50% of the whole sample to collect.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >18 years old with a diagnosis of non-dialysis chronic kidney disease at stage 2, 3 and 4.
2. Adult patients >18 years old with a diagnosis of end stage renal disease "stage 5".
3. Recorded data of Glomerular Filtration Rate for every patient.
4. Recorded data for dialysis patients (HCV, platelets count, creatinine, blood urea nitrogen, urea level and partial thromboplastin time).

Exclusion Criteria:

1. Adult patients <18 years.
2. End stage renal disease undergoing peritoneal dialysis.
3. Patients not physically able to participate in oral examination.
4. Patients with kidney transplantation.
5. Patients undergoing renal dialysis for reasons other than chronic kidney disease, such as acute renal failure, accidents, trauma, snake poisoning.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A convenience sample of adult patients diagnosed with chronic kidney disease attending at the Nephrology units at El Kasr Al-Ainy Cairo University Hospital will be enrolled in the study in a consecutive order
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Primary Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
oral mucosal lesion | 10 minutes
  Clinical examination according to WHO guidelines

SECONDARY OUTCOMES:
.Periodontal condition | 10 minutes
  Basic periodontal examination
Hepatitis C Virus at dialysis stage | 5 minutes
  HCV antibodies in patient blood

CONTACTS AND LOCATIONS:
Overall Officials: Mariam fakhr, Study Chair — the Nephrology units at the Kasr Al-Ainy Cairo university hospital.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gautam NR, Gautam NS, Rao TH, Koganti R, Agarwal R, Alamanda M. Effect of end-stage renal disease on oral health in patients undergoing renal dialysis: A cross-sectional study. J Int Soc Prev Community Dent. 2014 Sep;4(3):164-9. doi: 10.4103/2231-0762.142006. PMID 25374834